CLINICAL TRIAL: NCT03551730
Title: A Randomized, Double-blind, Vehicle-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Intravenously Administered PRT064445 After Dosing to Steady State With One of Four Direct/Indirect Factor Xa (fXa) Inhibitors in Healthy Volunteers.
Brief Title: Phase 2 Healthy Volunteer Study to Evaluate the Ability of PRT064445 to Reverse the Effects of Several Blood Thinner Drugs on Laboratory Tests (Module 3 of 4)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-502 Module 3
Record Dates: First submitted 2018-05-15; First posted 2018-06-11 (Actual); Results first posted 2018-08-13 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — PRT064445; Enoxaparin

STUDY DESIGN:
Intervention Model Description: This study has four modules with a total of 21 cohorts, each module was reported and submitted separately.
  Module 1, NCT01758432 (54 subjects with 7 cohorts including placebo); Module 2, NCT03578146 (48 subjects with 6 cohorts including placebo); Module 3, NCT03551730 (27 subjects with 4 cohorts including placebo); Module 4, NCT03551743 (28 subjects with 4 cohorts including placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Module 3 (210 mg bolus) original (Experimental): 210 mg PRT064445 given as a single IV bolus
  Interventions: Combination Product: PRT064445/Enoxaparin; Combination Product: Placebo/Enoxaparin
- Module 3 (420 mg bolus) original (Experimental): 420 mg PRT064445 given as a single IV bolus
  Interventions: Combination Product: PRT064445/Enoxaparin; Combination Product: Placebo/Enoxaparin
- Module 3 (210 mg) lyophilized (Experimental): 210 mg PRT064445 (lyophilized formulation) given as a single IV bolus
  Interventions: Combination Product: PRT064445/Enoxaparin; Combination Product: Placebo/Enoxaparin
- Module 3 Placebo (Placebo Comparator): Placebo administered intravenously (IV) as a bolus.
  Interventions: Drug: Placebo

INTERVENTIONS:
Combination Product: PRT064445/Enoxaparin
  Other Names: Andexanet
  Arms: Module 3 (210 mg bolus) original; Module 3 (210 mg) lyophilized; Module 3 (420 mg bolus) original
Combination Product: Placebo/Enoxaparin
  Arms: Module 3 (210 mg bolus) original; Module 3 (210 mg) lyophilized; Module 3 (420 mg bolus) original
Drug: Placebo
  Arms: Module 3 Placebo

SUMMARY:
The purpose of this study is to evaluate the ability of PRT064445 to reverse the effects of several blood thinner drugs on laboratory tests. The study also is evaluating the blood levels of PRT064445 given at different doses.

DETAILED DESCRIPTION:
A randomized, double-blind, vehicle-controlled study to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of intravenously administered PRT064445 after dosing to steady state with one of four direct/indirect factor Xa (fXa) inhibitors in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women between the ages of 18 and 45 years old

Exclusion Criteria:

* History (including family history) or symptoms of, or risk factors for bleeding
* History (including family history) of or risk factors for a hypercoagulable or thrombotic condition
* Absolute/relative contraindication to anticoagulation or treatment with specific anticoagulants
* History of major surgery, severe trauma or bone fracture within 3 months prior to dosing; or planned surgery within 1 month after dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tempe, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred at investigative site in the US between August 2013 through November 2013
Pre-assignment Details: Enoxaparin was administered subcutaneously at 40 mg once daily for 6 days to steady-state in an open label fashion. Subjects were then randomized to receive study treatment intravenously on Day 6; such that they ended at 3 hours after the last dose of enoxaparin.
Groups:
- Placebo: Placebo administered intravenously (IV) as a bolus.
- Module 3 (210 mg Bolus) Original; Module 3 (210 mg) Lyophilized: 210 mg andexanet IV bolus over 7 minutes (~30 mg/min)
- Module 3 (420 mg Bolus) Original: 420 mg andexanet IV bolus over 14 minutes (~30 mg/min)
Period: Overall Study
Arm/Group | Placebo | Module 3 (210 mg Bolus) Original | Module 3 (420 mg Bolus) Original | Module 3 (210 mg) Lyophilized
Started | 9 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 27 subjects were enrolled in Module 3
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Module 3 (210 mg Bolus) Original | Module 3 (420 mg Bolus) Original | Module 3 (210 mg) Lyophilized | Total
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (5.59) | 33.2 (8.30) | 32.5 (5.09) | 35.7 (8.66) | 33.7 (6.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 0 | 3 | 10
  Male | 4 | 4 | 6 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Efficacy:Percent Change From Baseline in Anti-fXa Activity at 2 Mins Following Andexanet/Placebo Administration Activity
Description: Anti-fXa activity was measured immediately prior to (Baseline) and at 2 mins following andexanet/placebo administration. Anti-fXa activity was measured using a commercial kit (Coamatic Heparin-82 33 9363, DiaPharma)
Time Frame: Baseline to 2 minutes following the end of andexanet/placebo administration
Population: 26 subjects who received andexanet or placebo were included in the pharmacodynamics (PD) analysis
Measure: Mean (Standard Deviation); unit: Percent change in anti-fXa activity
Arm/Group | Placebo | Module 3 (210 mg Bolus) Original | Module 3 (420 mg Bolus) Original | Module 3 (210 mg) Lyophilized
Number analyzed (Participants) | 8 | 6 | 6 | 6
Percent change in anti-fXa activity | -3.57 (12.80) | -70.80 (6.98) | -60.83 (8.39) | -69.85 (7.46)
Statistical Analysis 1: Comparison: Placebo vs Module 3 (210 mg Bolus) Original; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -0.23
Statistical Analysis 2: Comparison: Placebo vs Module 3 (420 mg Bolus) Original; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -0.20
Statistical Analysis 3: Comparison: Placebo vs Module 3 (210 mg) Lyophilized; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -0.23

2. Secondary Outcome: Efficacy: Percent Change From Baseline in Thrombin Generation at 2 Mins Following Andexanet/Placebo Administration
Description: Thrombin generation was measured immediately prior to (Baseline) and at 2 mins following andexanet/placebo administration. Thrombin generation was measured using a TF-initiated thrombin generation assay.
Time Frame: Baseline to 2 minutes following the end of andexanet/placebo administration
Population: 26 subjects who received andexanet or placebo were included in the PD analysis
Measure: Mean (Standard Deviation); unit: Percent change in thrombin generation
Arm/Group | Placebo | Module 3 (210 mg Bolus) Original | Module 3 (420 mg Bolus) Original | Module 3 (210 mg) Lyophilized
Number analyzed (Participants) | 8 | 6 | 6 | 6
Percent change in thrombin generation | 3.48 (15.162) | 36.34 (15.127) | 107.48 (73.301) | 72.7 (74.301)
Statistical Analysis 1: Comparison: Placebo vs Module 3 (210 mg Bolus) Original; Test type: Superiority; p = 0.1529, ANCOVA; Least Squares Means (Difference) = 53922.58
Statistical Analysis 2: Comparison: Placebo vs Module 3 (420 mg Bolus) Original; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = 124993.1
Statistical Analysis 3: Comparison: Placebo vs Module 3 (210 mg) Lyophilized; Test type: Superiority; p = 0.0032, ANCOVA; Least Squares Means (Difference) = 96385.09

3. Secondary Outcome: Andexanet Maximum Observed Plasma Concentration (Cmax)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. Cmax was taken directly from the raw data.
Time Frame: Blood was collected at predose, 0.033, 0.2, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4.5, 5.5, 6.5, 7.5, 8.5 and 14.5 hours postdose.
Population: 18 subjects who received andexanet were included in the andexanet pharmacokinetics (PK) analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Module 3 (210 mg Bolus) Original | Module 3 (420 mg Bolus) Original | Module 3 (210 mg) Lyophilized
Number analyzed (Participants) | 0 | 6 | 6 | 6
ng/mL |  | 32000 (7320) | 55800 (6050) | 42700 (14400)

4. Secondary Outcome: Andexanet Area Under the Drug Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf )
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. AUC0-inf was calculated using a non-compartmental approach
Time Frame: as for outcome 3
Population: 18 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Placebo | Module 3 (210 mg Bolus) Original | Module 3 (420 mg Bolus) Original | Module 3 (210 mg) Lyophilized
Number analyzed (Participants) | 0 | 6 | 6 | 6
ng*hr/mL |  | 33600 (4280) | 63900 (8880) | 40900 (12300)

5. Secondary Outcome: Andexanet Time of Maximum Observed Plasma Concentration (Tmax)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. Tmax was taken directly from the raw data.
Time Frame: as for outcome 3
Population: 18 subjects who received andexanet were included in the andexanet PK analysis
Measure: Median (Full Range); unit: hr
Arm/Group | Placebo | Module 3 (210 mg Bolus) Original | Module 3 (420 mg Bolus) Original | Module 3 (210 mg) Lyophilized
Number analyzed (Participants) | 0 | 6 | 6 | 6
hr |  | 0.18 [0.16 to 0.35] | 0.29 [0.27 to 0.54] | 0.17 [0.17 to 0.19]

6. Secondary Outcome: Andexanet Apparent Terminal Elimination Half-life (t1/2)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay.t1/2 was determined by linear regression of the log concentration on the terminal portion of the plasma concentration-time curve.
Time Frame: as for outcome 3
Population: 18 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Placebo | Module 3 (210 mg Bolus) Original | Module 3 (420 mg Bolus) Original | Module 3 (210 mg) Lyophilized
Number analyzed (Participants) | 0 | 6 | 6 | 6
hr |  | 5.28 (1.99) | 6.11 (2.34) | 8.36 (7.46)

7. Secondary Outcome: Andexanet Total Systemic Clearance (CL)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. CL was calculated using a non-compartmental approach.
Time Frame: as for outcome 3
Population: 18 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Placebo | Module 3 (210 mg Bolus) Original | Module 3 (420 mg Bolus) Original | Module 3 (210 mg) Lyophilized
Number analyzed (Participants) | 0 | 6 | 6 | 6
L/hr |  | 6.34 (0.870) | 6.69 (0.991) | 5.56 (1.76)

8. Secondary Outcome: Andexanet Total Volume of Distribution (Vss)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. Vss was calculated using a non-compartmental approach.
Time Frame: as for outcome 3
Population: 18 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Placebo | Module 3 (210 mg Bolus) Original | Module 3 (420 mg Bolus) Original | Module 3 (210 mg) Lyophilized
Number analyzed (Participants) | 0 | 6 | 6 | 6
L |  | 9.86 (2.61) | 9.62 (1.13) | 9.69 (4.16)

ADVERSE EVENTS:
Time Frame: ~7 weeks
Description: Only subjects who received at least one dose of study drug were included in the safety analysis.
Groups:
- Placebo: Placebo was administered intravenously (IV) as a bolus
- Module 3 (210 mg Andexanet) Original Formulation: 210 mg andexanet IV bolus over 7 minutes (~30 mg/min)
- Module 3 (420 mg Andexanet) Original Forumulation: 420 mg andexanet IV bolus over 14 minutes (~30 mg/min) 420 mg andexanet IV bolus over 14 minutes (~30 mg/min)
- Module 3 (210 mg Andexanet ) Lyophilized: 210 mg andexanet IV bolus over 7 minutes (~30 mg/min) 210 mg andexanet IV bolus over 7 minutes (~30 mg/min)
Arm/Group | Placebo | Module 3 (210 mg Andexanet) Original Formulation | Module 3 (420 mg Andexanet) Original Forumulation | Module 3 (210 mg Andexanet ) Lyophilized
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/8 | 4/6 | 4/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Module 3 (210 mg Andexanet) Original Formulation (N=6) | Module 3 (420 mg Andexanet) Original Forumulation (N=6) | Module 3 (210 mg Andexanet ) Lyophilized (N=6)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural hematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Conducted in healthy volunteers at Clinical Research Organization